CLINICAL TRIAL: NCT04033926
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Crossover Multicenter Study to Evaluate the Safety and Efficacy of KZR-616 in the Treatment of Patients With Active Polymyositis or Dermatomyositis
Brief Title: A Phase 2 Study of KZR-616 to Evaluate Safety and Efficacy in Patients With Active Polymyositis or Dermatomyositis
Acronym: PRESIDIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KZR-616-003
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: Myositis; Idiopathic inflammatory myopathies; Polymyositis; Dermatomyositis; Musculoskeletal Diseases; Muscular Diseases
MeSH Terms: conditions — Polymyositis; Dermatomyositis; Myositis; Musculoskeletal Diseases; Muscular Diseases | interventions — KZR-616

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): * Treatment Period 1: KZR-616 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
  * Treatment Period 2: Placebo SC weekly for 16 weeks
  Interventions: Drug: KZR-616; Drug: Placebo
- Arm B (Other): * Treatment Period 1: Placebo SC weekly for 16 weeks
  * Treatment Period 2: KZR-616 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
  Interventions: Drug: KZR-616; Drug: Placebo

INTERVENTIONS:
Drug: KZR-616 — Subcutaneous 30 mg weekly for 2 weeks, then 45 mg weekly for 14 weeks
  Other Names: zetomipzomib
Drug: Placebo — Subcutaneous injection for 16 weeks

SUMMARY:
This was a Phase 2 randomized, double-blind, placebo-controlled, crossover, multicenter study to evaluate the safety, tolerability, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of treatment with KZR-616 in patients with active polymyositis (PM) or dermatomyositis (DM). Patients were evaluated for eligibility during the Screening Period. Eligible patients were stratified by diagnosis of DM or PM and randomized 1:1 to Arm A or Arm B of the study.

During the 32-week treatment period, patients received study drug subcutaneously (SC) once weekly with 2 treatment periods of 16 weeks each.

This study was conducted on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients at least 18 years of age
2. Body Mass Index (BMI) of 18 to 40 kg/m^2
3. Diagnosis of probable or definite DM or PM by the 2017 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) Classification Criteria
4. Must have their data reviewed by an adjudication committee to confirm eligibility unless at least 1 of the following is present:

   1. Muscle biopsy with evidence of active myositis within the last 6 months prior to or at Screening
   2. Electromyography or magnetic resonance imaging with evidence of active myositis within the last 6 months prior to Screening
   3. A creatine kinase (CK) ≥4 × upper limit of normal (ULN).
5. Must have demonstrable muscle weakness as measured by the Manual Muscle Testing-8 muscle Groups (MMT-8) with a score ≥80/150 but ≤136/150 units and any 2 of the following:

   1. Physician Global Assessment (MDGA) visual analog scale (VAS) ≥2 cm
   2. Patient Global Assessment of Disease Activity (PtGADA) VAS ≥2 cm
   3. At least one muscle enzyme laboratory measurement ≥1.3 × ULN
   4. Myositis Disease Activity Assessment Tool (MDAAT) Extramuscular Global Activity VAS ≥1 cm.
6. Documented inadequate response OR have demonstrated documented toxicity or intolerance to prior standard of care therapies
7. Has had age-appropriate cancer screening that is up to date and negative for evidence of malignancy as per local standard of care

Exclusion Criteria:

1. Has significant muscle damage or has a muscle damage VAS score ≥5 cm on the MDI
2. Any other form of myositis or myopathy other than PM or DM
3. Any condition that precludes the ability to quantitate muscle strength
4. Has severe interstitial lung disease or has a pulmonary damage VAS score ≥5 cm on the Myositis Damage Index (MDI)
5. Presence of autoinflammatory disease
6. Use of nonpermitted medications or treatments within the specified washout periods prior to screening
7. Patient has had recent serious or ongoing infection, or risk for serious infection
8. Any of the following laboratory values at Screening:

   1. Estimated glomerular filtration rate <45 mL/min
   2. Hemoglobin <10 g/dL
   3. White blood cell (WBC) count <3.0 × 10^9/L
   4. Absolute neutrophil count (ANC) <1.5 × 10^9/L (1500/mm^3)
   5. Platelet count <100 × 10^9/L
   6. Serum AST or serum ALT >2.5 × ULN (unless considered consistent with muscle origin)
   7. Serum alkaline phosphatase >2.5 × ULN
   8. Total bilirubin >1.5 × ULN (3 × ULN for patients with documented Gilbert's syndrome)
   9. Thyroid stimulating hormone outside of the central laboratory normal range
   10. Immunoglobulin G (IgG) <500 mg/dL.
9. Presence of New York Heart Association Class III or IV heart failure, or uncontrolled blood pressure, or prolonged QT interval
10. Major surgery within 12 weeks before Screening or planned during the study period
11. Clinical evidence of significant unstable or uncontrolled diseases
12. Any active or suspected malignancy, including myeloproliferative or lymphoproliferative disorder, or history of documented malignancy within the last 5 years before Screening or within 3 years of diagnosis of myositis, except appropriately excised and cured cervical carcinoma in situ or basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kezar, Study Director — Kezar Life Sciences, Inc.
Locations (14):
- United States (12):
  - KZR Research Site, Beverly Hills, California
  - KZR Research Site, Orange, California
  - KZR Research Site, Miami, Florida
  - KZR Research Site, Atlanta, Georgia
  - KZR Research Site, Kansas City, Kansas
  - KZR Research Site, Baltimore, Maryland
  - KZR Research Site, Ann Arbor, Michigan
  - KZR Research Site, Great Neck, New York
  - KZR Research Site, Duncansville, Pennsylvania
  - KZR Research Site, Pittsburgh, Pennsylvania
  - KZR Research Site, Austin, Texas
  - KZR Research Site, Henrico, Virginia
- KZR Research Site, Prague, Czechia
- KZR Research Site, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had a cross-over design. There was a 32-week double-blind Treatment Period divided into two 16-week treatment periods. Participants enrolled at the end of Treatment Period 2 were allowed to join an optional open-label extension study, KZR-616-003E (NCT04628936).
Groups:
- Zetomipzomib First, Then Placebo (Arm A): Treatment Period 1: Zetomipzomib 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
  Treatment Period 2: Placebo SC weekly for 16 weeks
- Placebo First, Then Zetomipzomib (Arm B): Treatment Period 1: Placebo SC weekly for 16 weeks
  Treatment Period 2: Zetomipzomib 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
Period: Treatment Period 1
Arm/Group | Zetomipzomib First, Then Placebo (Arm A) | Placebo First, Then Zetomipzomib (Arm B)
Started | 13 | 12
Completed | 10 | 12
Not Completed | 3 | 0
Period: Treatment Period 2
Arm/Group | Zetomipzomib First, Then Placebo (Arm A) | Placebo First, Then Zetomipzomib (Arm B)
Started | 10 | 12
Completed | 8 | 12
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zetomipzomib First, Then Placebo (Arm A): * Treatment Period 1: Zetomipzomib 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
  * Treatment Period 2: Placebo SC weekly for 16 weeks
- Placebo First, Then Zetomipzomib (Arm B): * Treatment Period 1: Placebo SC weekly for 16 weeks
  * Treatment Period 2: Zetomipzomib 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
- Total: Total of all reporting groups
Arm/Group | Zetomipzomib First, Then Placebo (Arm A) | Placebo First, Then Zetomipzomib (Arm B) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.7) | 54.3 (16.4) | 51.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Physician Global Assessment (MDGA) [Mean (Standard Deviation); unit: score on a scale] — One of the International Myositis Assessment and Clinical Studies Group (IMACS) core set activity measures (CSAMs). The Physician Global Assessment (MDGA) is a physician assessment of the patient's overall disease activity at the time of the assessment. The responses range from none/no evidence of disease activity to extremely active/severe disease activity on a scale of 0 to 10. Higher numbers represent more severe disease activity.
  score on a scale | 5.1 (1.3) | 4.9 (1.6) | 5.0 (1.4)
Patient Global Assessment of Disease Activity (PtGADA) [Mean (Standard Deviation); unit: score on a scale] — One of the IMACS CSAMs. The Patient Global Assessment of Disease Activity (PtGADA) is a patient assessment of their overall disease activity at the time of the assessment. The responses range from no evidence of disease activity to severe disease activity on a scale of 0 to 100. Higher numbers represent more severe disease activity.
  score on a scale | 68.8 (20.5) | 58.6 (18.9) | 63.9 (20.0)
Manual Muscle Testing-8 Muscle Groups (MMT-8) [Mean (Standard Deviation); unit: score on a scale] — One of the IMACS CSAMs. The Manual Muscle Testing-8 Muscle Groups (MMT-8) scores range from 0-150, where higher scores represent more muscle strength.
  score on a scale | 124.2 (9.5) | 127.7 (6.5) | 125.9 (8.2)
Health Assessment Questionnaire - Disability (HAQ-DI) [Mean (Standard Deviation); unit: score on a scale] — One of the IMACS CSAMs. The Health Assessment Questionnaire - Disability (HAQ-DI) scores range from 0-3, where higher scores represent less physical function.
  score on a scale | 1.7 (0.9) | 1.2 (0.7) | 1.5 (0.8)
The Extramuscular Global Assessment of the Myositis Disease Activity Assessment Tool (MDAAT) [Mean (Standard Deviation); unit: score on a scale] — One of the IMACS CSAMs. The Extramuscular Global Assessment of the Myositis Disease Activity Assessment Tool (MDAAT) (2005 version) scores range from 0 - 10, where higher scores represent more disease activity outside of muscle.
  score on a scale | 2.3 (1.9) | 2.8 (2.4) | 2.5 (2.1)
Muscle Enzymes [Mean (Standard Deviation); unit: U/L] — One of the IMACS CSAMs. Muscle enzymes summarize the most abnormal clinical laboratory assessment (creatine kinase [CK], aldolase, lactate dehydrogenase [LDH], alanine aminotransferase [ALT], or aspartate aminotransferase [AST]) at baseline; lower scores are better and indicate less muscle damage.
  U/L | 2752.7 (4521.1) | 2070.4 (3108.2) | 2425.2 (3843.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Total Improvement Score (TIS) From Start to End of Zetomipzomib (KZR-616) Treatment Period
Description: The primary efficacy endpoint was mean change from start to end of zetomipzomib (KZR-616) Treatment Periods in the Total Improvement Score (TIS), which ranges from 0 to 100 [low of 0 to high of 100, where higher scores are better]. Mean change in TIS was calculated by comparing the Baseline and post Baseline observations for patients in both KZR-616 treatment periods combined.
  Note: TIS scores for placebo treatment periods are presented in this outcome measure but were not included in the primary outcome measure analysis.
Time Frame: 16 weeks in each Treatment Period (32 weeks total)
Population: For the first 16 weeks, analysis was done for Treatment Period 1. For the second 16 weeks, analysis was done for Treatment Period 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm A: Period 1 (Zetomipzomib); Arm B: Period 2 (Zetomipzomib): Zetomipzomib 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
- Arm B: Period 1 (Placebo); Arm A: Period 2 (Placebo): Placebo SC weekly for 16 weeks
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm B: Period 1 (Placebo) | Arm A: Period 2 (Placebo) | Arm B: Period 2 (Zetomipzomib)
Number analyzed (Participants) | 10 | 12 | 8 | 12
score on a scale | 25.5 (18.6) | 25.0 (19.9) | 33.1 (17.6) | 33.5 (22.9)

2. Secondary Outcome: Proportion of Patients With TIS Response
Description: The proportion of patients with an increase of ≥ 20 points on the TIS from start to end of zetomipzomib (KZR-616) treatment. TIS response is categorized by the following improvement thresholds:
  * Minimal response = TIS ≥ 20
  * Moderate response = TIS ≥ 40
  * Major response = TIS ≥ 60
  This endpoint was assessed by comparing Week 16 versus Week 0 for patients allocated to Arm A and Week 32 versus Week 16 for patients allocated to Arm B. This re-baselining approach was utilized to maximize the precision for assessment of zetomipzomib effect in Arm B.
Time Frame: 16 weeks in each Treatment Period (32 weeks total)
Measure: Number; unit: participants
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm B: Period 1 (Placebo) | Arm A: Period 2 (Placebo) | Arm B: Period 2 (Zetomipzomib)
Number analyzed (Participants) | 10 | 12 | 8 | 12
participants
  Minimal (TIS ≥ 20) | 6 | 7 | 1 | 6
  Moderate (TIS ≥ 40) | 2 | 2 | 1 | 2
  Major (TIS ≥ 60) | 0 | 1 | 0 | 1

3. Secondary Outcome: Number of Patients Meeting the International Myositis Assessment and Clinical Studies Group (IMACS) Definition of Improvement (DOI)
Description: The IMACS DOI is ≥ 20% improvement in at least 3 of 6 core set activity measures, with no more than 2 core set activity measures (CSAMs) worsening by ≥ 25% (Manual Muscle Testing-8 Muscle Groups [MMT-8] could not be a worsening measure).
Time Frame: 16 weeks in each Treatment Period (32 weeks total)
Measure: Number; unit: participants
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm B: Period 1 (Placebo) | Arm A: Period 2 (Placebo) | Arm B: Period 2 (Zetomipzomib)
Number analyzed (Participants) | 13 | 12 | 10 | 12
participants | 1 | 1 | 1 | 3

4. Secondary Outcome: Mean Percent Change From Baseline From Start to End of Treatment in the IMACS Individual CSAMs
Description: Mean percent change from baseline of the IMACS CSAMs consisting of:
  * Physician Global Assessment: physician assessment of patient's overall disease activity at present, high numbers indicate more severe disease activity [0-10]
  * Patient Global Assessments of Disease Activity: patient assessment of their overall disease activity at present, high numbers indicate more severe disease activity [0-100]
  * Manual Muscle Testing-8 Muscle Groups: scores range from 0 - 150, high scores are better
  * Health Assessment Questionnaire-Disability Index: scores range from 0 - 3, high scores are worse
  * Extramuscular Global Assessment of the Myositis Disease Activity Assessment Tool (2005 version): scores range from 0 - 10, high scores are worse
  * Muscle enzymes (clinical laboratory assessments [CLA]): Summarize the most abnormal CLA (creatine kinase [CK], aldolase, lactate dehydrogenase [LDH], alanine aminotransferase [ALT], or aspartate aminotransferase [AST]) at baseline, lower scores are better
Time Frame: 16 weeks in each Treatment Period (32 weeks total)
Population: Some values were not collected for participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm B: Period 1 (Placebo) | Arm A: Period 2 (Placebo) | Arm B: Period 2 (Zetomipzomib)
Number analyzed (Participants) | 10 | 12 | 8 | 12
percent change
  Physician Global Assessment (MDGA) | -32.5 (35.1) | -22.1 (36.8) | 81.7 (204.3) | -4.5 (58.6)
  Patient Global Assessments of Disease Activity (PtGADA): number analyzed (Participants) | 8 | 11 | 8 | 10
  Patient Global Assessments of Disease Activity (PtGADA) | -23.1 (35.1) | -21.7 (49.8) | 48.6 (121.4) | 64.4 (163.8)
  Manual Muscle Testing-8 Muscle Groups (MMT-8) | 6.7 (8.6) | 5.6 (6.1) | 0.2 (4.6) | 1.5 (7.1)
  Health Assessment Questionnaire-Disability Index (HAQ-DI): number analyzed (Participants) | 7 | 11 | 7 | 9
  Health Assessment Questionnaire-Disability Index (HAQ-DI) | -28.2 (34.4) | 1.2 (80.5) | 19.2 (51.2) | -8.8 (60.4)
  The Extramuscular Global Assessment of the Myositis Disease Activity Assessment Tool (MDAAT): number analyzed (Participants) | 9 | 11 | 8 | 10
  The Extramuscular Global Assessment of the Myositis Disease Activity Assessment Tool (MDAAT) | -14.6 (75.2) | -14.7 (68.7) | 0.8 (69.4) | -34.8 (47.5)
  Muscle enzymes (clinical laboratory assessments) | -19.8 (24.1) | 8.7 (44.2) | -3.9 (42.6) | -8.3 (50.6)

5. Secondary Outcome: Mean Change in CDASI From Start to End of Zetomipzomib (KZR-616) Treatment
Description: Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) is a clinician scored single-page instrument that separately measures activity and damage, which consists of three (3) activity measures and two (2) damage measures which are assessed over 15 body areas. Scores range from 0-100 for activity and from 0-32 for damage, with higher scores indicating more severe disease.
Time Frame: 16 weeks in each Treatment Period (32 weeks total)
Population: This measure was only performed for patients with DM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm B: Period 1 (Placebo) | Arm A: Period 2 (Placebo) | Arm B: Period 2 (Zetomipzomib)
Number analyzed (Participants) | 5 | 6 | 5 | 6
score on a scale
  Activity Score | -2.2 (5.3) | -1.2 (13.5) | -4.4 (5.2) | -0.2 (16.1)
  Damage Score | 0.0 (0.7) | -0.8 (2.1) | -0.2 (0.8) | -1.7 (3.1)

6. Secondary Outcome: Mean Change in PP-NRS From Start to End of Zetomipzomib (KZR-616) Treatment
Description: The Peak Pruritus Numeric Rating Scale (PP-NRS) is used to evaluate severity of itch in DM patients. Scores range from 0-10, with zero (0) representing no itch and ten (10) representing the worst itch imaginable within a 24-hour recall period.
Time Frame: 16 weeks in each Treatment Period (32 weeks total)
Population: This measure was only performed for patients with DM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm B: Period 1 (Placebo) | Arm A: Period 2 (Placebo) | Arm B: Period 2 (Zetomipzomib)
Number analyzed (Participants) | 5 | 6 | 5 | 6
score on a scale | -1.8 (1.3) | -2.0 (4.2) | -2.0 (1.9) | -3.5 (3.5)

7. Secondary Outcome: PK of Zetomipzomib [KZR-616] (Cmax)
Description: This is the maximum observed plasma concentration (Cmax) observed after administration of the first dose of KZR-616 (either Week 0 or Week 16). The pharmacokinetic (PK) parameters were calculated using all timepoints at which the concentration was measured, ie. pre-dose and 30 minutes, and 4 hours post-dose, with an additional sample obtained at 0.25, 1, or 2 hours post-dose.
Time Frame: Up to 5 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Zetomipzomib (Arm A: Period 1); Zetomipzomib (Arm B: Period 2): Zetomipzomib 30 mg SC weekly for 2 weeks, then 45 mg SC weekly for 14 weeks
Arm/Group | Zetomipzomib (Arm A: Period 1) | Zetomipzomib (Arm B: Period 2)
Number analyzed (Participants) | 13 | 12
ng/mL | 57.5 (78.9) | 82.3 (42.5)

8. Secondary Outcome: PK of Zetomipzomib [KZR-616] (Tmax)
Description: This is the time to maximum observed plasma concentration (tmax) observed after administration of the first dose of KZR-616 (either Week 0 or Week 16). The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 30 minutes, and 4 hours postdose, with an additional sample obtained at 0.25, 1, or 2 hours postdose.
Time Frame: Up to 5 hours
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Zetomipzomib (Arm A: Period 1) | Zetomipzomib (Arm B: Period 2)
Number analyzed (Participants) | 13 | 12
hours | 0.50 [0.25 to 0.53] | 0.50 [0.25 to 0.55]

9. Secondary Outcome: PK of Zetomipzomib [KZR-616] (AUC)
Description: This is the area under the curve (AUC) from predose through 4 hour postdose observed after administration of the first dose of KZR-616 (either Week 0 or Week 16). The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 30 minutes, and 4 hours postdose, with an additional sample obtained at 0.25, 1, or 2 hours postdose.
Time Frame: Up to 5 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Zetomipzomib (Arm A: Period 1) | Zetomipzomib (Arm B: Period 2)
Number analyzed (Participants) | 12 | 12
ng*h/mL | 120 (59.0) | 156 (40.4)

10. Secondary Outcome: PK of KZR-59587 (Cmax)
Description: This is the maximum observed plasma concentration of KZR-59587 (Cmax) observed after administration of the first dose of KZR-616 (either Week 0 or Week 16). The pharmacokinetic (PK) parameters were calculated using all timepoints at which the concentration was measured, ie. pre-dose and 30 minutes, and 4 hours post-dose, with an additional sample obtained at 0.25, 1, or 2 hours post-dose.
Time Frame: Up to 5 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Zetomipzomib (Arm A: Period 1) | Zetomipzomib (Arm B: Period 2)
Number analyzed (Participants) | 13 | 12
ng/mL | 48.2 (58.5) | 58.5 (46.4)

11. Secondary Outcome: PK of KZR-59587 (Tmax)
Description: This is the time to maximum observed plasma concentration of KZR-59587 (tmax) observed after administration of the first dose of KZR-616 (either Week 0 or Week 16). The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 30 minutes, and 4 hours postdose, with an additional sample obtained at 0.25, 1, or 2 hours postdose.
Time Frame: Up to 5 hours
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Zetomipzomib (Arm A: Period 1) | Zetomipzomib (Arm B: Period 2)
Number analyzed (Participants) | 13 | 12
hours | 2.50 [0.52 to 4.02] | 3.92 [0.98 to 4.55]

12. Secondary Outcome: PK of KZR-59587 (AUC)
Description: This is the area under the curve of KZR-59587 (AUC) from predose through 4 hour postdose observed after administration of the first dose of KZR-616 (either Week 0 or Week 16). The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose and 30 minutes, and 4 hours postdose, with an additional sample obtained at 0.25, 1, or 2 hours postdose.
Time Frame: Up to 5 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Zetomipzomib (Arm A: Period 1) | Zetomipzomib (Arm B: Period 2)
Number analyzed (Participants) | 12 | 12
ng*h/mL | 150 (59.2) | 176 (53.3)

ADVERSE EVENTS:
Time Frame: Up to 40 weeks
Arm/Group | Arm A: Period 1 (Zetomipzomib) | Arm A: Period 2 (Placebo) | Arm B: Period 1 (Placebo) | Arm B: Period 2 (Zetomipzomib)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/10 | 1/12 | 1/12
Other Adverse Events (participants affected / at risk) | 12/13 | 8/10 | 7/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Period 1 (Zetomipzomib) (N=13) | Arm A: Period 2 (Placebo) (N=10) | Arm B: Period 1 (Placebo) (N=12) | Arm B: Period 2 (Zetomipzomib) (N=12)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Period 1 (Zetomipzomib) (N=13) | Arm A: Period 2 (Placebo) (N=10) | Arm B: Period 1 (Placebo) (N=12) | Arm B: Period 2 (Zetomipzomib) (N=12)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (7) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (12) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (40) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (7) | 1 (1) | 0 (0) | 2 (14)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 5 (13) | 0 (0) | 0 (0) | 2 (25)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 6 (32) | 0 (0) | 1 (2) | 2 (2)
Injection site pruritus (General disorders) | 2 (9) | 0 (0) | 0 (0) | 1 (9)
Injection site rash (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 3 (31) | 0 (0) | 2 (4) | 6 (57)
Injection site streaking (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site swelling (General disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (24) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (17) | 0 (0) | 0 (0) | 1 (3)
Vaccination site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema migrans (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Post procedural pruritus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biopsy (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dizziness exertional (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (13) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mechanic's hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (2) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
* This study was not powered to detect statistical differences between treatment arms.
* Crossover study design with no washout period may have confounded assessments.
* Limited information from the safety follow-up as most patients elected to join the OLE study (NCT04628936).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall have the right to publish or present their own data resulting from the Study ("Publication") upon the earlier of: (a) the date following a multicenter publication coordinated by Sponsor regarding the Protocol; (b) 12 months after completion of the Protocol by all sites; or (c) the date after submission of the Study Data by Sponsor to the FDA.

The PI must furnish Sponsor with a copy of any Publication at least 30 days in advance of the proposed submission or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04033926/Prot_SAP_000.pdf